CLINICAL TRIAL: NCT06203210
Title: A Phase 3, Multicenter, Randomized, Open-label Study of Ifinatamab Deruxtecan (I-DXd), a B7-H3 Antibody Drug Conjugate (ADC), Versus Treatment of Physician's Choice (TPC) in Subjects With Relapsed Small Cell Lung Cancer (SCLC) (IDeate-Lung02)
Brief Title: A Study of Ifinatamab Deruxtecan Versus Treatment of Physician's Choice in Subjects With Relapsed Small Cell Lung Cancer
Acronym: IDeate-Lung02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-188; 2023-509628-16-00 (Other: EU CT); 2031230631 (Other: jRCT)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; Ifinatamab deruxtecan; I-DXd
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; amrubicin; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifinatamab deruxtecan (I-DXd) (Experimental): Participants randomized to receive 12 mg/kg I-DXd monotherapy on Day 1 of each 21-day cycle until unacceptable toxicity, progressive disease (PD), or withdrawal of consent as specified in the protocol.
  Interventions: Drug: Ifinatamab deruxtecan
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants randomized to receive topotecan, lurbinectedin, or amrubicin, as per investigator's choice and per locally approved label (indicated dose and frequency), until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: Topotecan; Drug: Amrubicin; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Ifinatamab deruxtecan — 12 mg/kg intravenous dose on Day 1 of each 21-day cycle
  Other Names: I-DXd
  Arms: Ifinatamab deruxtecan (I-DXd)
Drug: Topotecan — Topotecan will be administered per local SoC.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Amrubicin — Amrubicin will be administered per local SoC.
  Arms: Treatment of Physician's Choice (TPC)
Drug: Lurbinectedin — Lurbinectedin will be administered per local SoC
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
This study was designed to compare the efficacy and safety of I-DXd with treatment of physician's choice in participants with relapsed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether treatment with I-DXd improves objective response rate (ORR) and prolongs overall survival (OS) compared with treatment of physician's choice among participants with relapsed SCLC.

The secondary objectives of the study are to further evaluate the efficacy/safety of I-DXd, health economics and outcome research measures (including patient reported outcomes), immunogenicity of I-DXd, B7-H3 protein expression, and characterize the pharmacokinetics of I-DXd.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all the following criteria to be eligible for randomization into the study:

1. Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
2. Adults ≥18 years or the minimum legal adult age (whichever is greater) at the time the informed consent form is signed.
3. Has histologically or cytologically documented extensive-stage small cell lung cancer (ES-SCLC).
4. The participant must provide adequate baseline tumor samples with sufficient quantity and quality of tumor tissue content.
5. Has received prior therapy with only one prior platinum-based line as systemic therapy for SCLC with at least 2 cycles of therapy and a chemotherapy free-interval of ≥30 days.
6. Has at least 1 measurable lesion according to RECIST v1.1 as assessed by the investigator.
7. Has documentation of radiological disease progression on or after the most recent systemic therapy.
8. Has ECOG PS of ≤1 within 7 days prior to Cycle 1 Day 1 (C1D1).
9. Has no evidence of brain or leptomeningeal disease (spinal cord or central nervous system [CNS] metastases) based on history and physical examination. Subjects must require no treatment with steroids or anticonvulsants and have a stable neurologic status for at least 2 weeks prior to the first dose of study drug.

Exclusion Criteria

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Has received prior treatment with orlotamab, enoblituzumab, or other B7 homologue 3 (B7-H3) targeted agents, including I-DXd.
2. Prior discontinuation of an antibody drug conjugate (ADC) that consists of an exatecan derivative (eg, trastuzumab deruxtecan) due to treatment-related toxicities.
3. Has received any of the comparators used in this study or any topoisomerase I inhibitor.
4. Has inadequate washout period before randomization as specified in the protocol.
5. Has any of the following conditions within the past 6 months: cerebrovascular accident, transient ischemic attack, or another arterial thromboembolic event.
6. Has uncontrolled or significant cardiovascular disease.
7. Has clinically significant corneal disease.
8. Has any history of ILD/pneumonitis irrespective of steroid use, or current ILD, or suspected ILD, or ILD that cannot be ruled out by imaging at Screening. Participants may be eligible if they had history of radiation pneumonitis that did not require steroids.

   Examples of suspected ILD/pneumonitis by imaging include the presence of lung parenchymal fibrosis, such as combined pulmonary fibrosis and emphysema (CPFE) and any radiographic features consistent with ILA, including but not limited to, extensive ground glass opacities, reticular opacities, traction bronchiectasis, and honeycombing.
9. Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses, including, but not limited to, any underlying pulmonary disorder and potential pulmonary involvement caused by any autoimmune, connective tissue, or inflammatory disorders, prior pneumonectomy, or requirement for supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Objective Response Rate Assessed by Blinded Independent Central Review | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on BICR by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Overall Survival | From the date of randomization to the date of death due to any cause, up to approximately 5 years

SECONDARY OUTCOMES:
Number of Participants With Objective Response Rate Assessed by Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on investigator by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Progression-free Survival As Assessed by Blinded Independent Central Review and Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  PFS is defined as the time interval from the date of randomization to the date of disease progression as per BICR and investigator assessment or death due to any cause.
Duration of Response As Assessed by Blinded Independent Central Review and Investigator | From the date of first documentation of confirmed response (CR or PR) to the first documentation of objective progression or to death due to any cause, whichever occurs first, up to approximately 5 years
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death. The DoR will be calculated for responding participants (PR or CR) only.
Disease Control Rate As Assessed by Blinded Independent Central Review and Investigator | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) by BICR and investigator assessment per RECIST v1.1.
Time to Response As Assessed by Blinded Independent Central Review and Investigator | From the start date of study drug to the date of the first documentation of response (CR or PR) that is subsequently confirmed, up to approximately 5 years
  TTR is defined as the time from the date of randomization to the first documentation of objective tumor response (CR or PR) that is subsequently confirmed by BICR and investigator assessment .Time to response (TTR) will be calculated for confirmed responders only.
Change from Baseline in The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 | Baseline up to 5 years
  This 30-item questionnaire assesses global health status (GHS)/quality of life (QoL), subject functioning, and general cancer symptoms and has a recall period of one week. All scores for the EORTC QLQ-C30 instrument are linearly transformed to a 0 to 100 metric, where a higher score on GHS/QoL and functioning scales indicates a better outcome and a higher score for the symptom scales indicates worse outcomes.
Change from Baseline in The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 29 (EORTC QLQ-LC29) | Baseline up to 5 years
  The LC29 is a self-reported 29-item questionnaire that measures SCLC-related symptoms and the side effects of treatments and has a recall period of one week. All scores range from 0 to 100, with a higher score indicating a worse outcome.
Overall Number of Participants With Treatment-emergent Adverse Events Following I-DXd Monotherapy | Baseline up to 5 years
  TEAEs are assessed based on NCI CTCAE v5.0.
The Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive At Any Time and Who Have A Treatment-emergent Anti-Drug Antibody | Baseline up to 5 years
  The ADA prevalence, which is the percentage of participants who are ADA positive at any time point (baseline or post-baseline), as well as the ADA incidence, which is the proportion of participants having treatment-emergent ADA during the study period, will only be reported in participants receiving I-DXd.
Pharmacokinetic Parameter Maximum Concentration for I-DXd, Total Anti-B7-H3 Antibody, and MAAA-1181a | Cycle 1 before infusion (BI), end of infusion EOI), and 3, 6, 24, 72, 168, 336, and 504 hours (hrs) post dose; Cycle 2 BI and EOI; Cycle 3 BI, EOI, and 6 hrs postdose; Cycles 4, 5, and every 2 cycles thereafter up to 5 years BI (each cycle is 21 days)
  Maximum concentration (Cmax) will be assessed using non-compartmental methods in participants randomized to the I-DXd group.
Pharmacokinetic Parameter Time to Maximum Concentration for I-DXd, Total Anti-B7-H3 Antibody, and MAAA-1181a | Cycle 1 before infusion (BI), end of infusion EOI), and 3, 6, 24, 72, 168, 336, and 504 hours (hrs) post dose; Cycle 2 BI and EOI; Cycle 3 BI, EOI, and 6 hrs postdose; Cycles 4, 5, and every 2 cycles thereafter up to 5 years BI (each cycle is 21 days)
  Time to maximum concentration (Tmax) will be assessed using non-compartmental methods in participants randomized to the I-DXd group.
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve for I-DXd, Total Anti-B7-H3 Antibody, and MAAA-1181a | Cycle 1 before infusion (BI), end of infusion EOI), and 3, 6, 24, 72, 168, 336, and 504 hours (hrs) post dose; Cycle 2 BI and EOI; Cycle 3 BI, EOI, and 6 hrs postdose; Cycles 4, 5, and every 2 cycles thereafter up to 5 years BI (each cycle is 21 days)
  Area under the plasma concentration-time curve up to the last quantifiable time point (AUClast) and area under the plasma concentration-time curve dosing interval (AUCtau) will be assessed using non-compartmental methods in participants randomized to the I-DXd group.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director, Study Director — Daiichi Sankyo
Locations (230):
- United States (29):
  - Highlands Oncology Group, Springdale, Arkansas
  - Clinical Research Providence Medical Foundation, Fullerton, California
  - UCLA Hematology-Oncology, Los Angeles, California
  - UCSF Mission Bay Mission Hall, San Francisco, California
  - University of Miami Hospital and Clinics Sylvester Comprehensive Cancer Center, Miami, Florida
  - AdventHealth Orlando, Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - John Hopkins School of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mercy Clinic Oncology and Hematology Sindelar Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Astera Cancer Care, East Brunswick, New Jersey
  - Meridian Health Systems, Neptune City, New Jersey
  - Clinical Research Alliance, Inc, Lake Success, New York
  - New York University Cancer Center - Laura and Isaac, New York, New York
  - Montefiore Medical Center Prime, The Bronx, New York
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Oncology/Hematology Care Clinical Trials, Llc, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - THE WEST CLINIC, PLLC dba West Cancer Center, Germantown, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
  - University of Texas Md Anderson Cancer Center, Houston, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Ballarat Base Hospital, Ballarat
  - Flinders Medical Centre (Fmc), Bedford Park
  - Chris O Brien Lifehouse, Camperdown
  - Sunshine Hospital, St Albans
  - St John of God Subiaco Hospital, Subiaco
  - Townsville Cancer Centre, Townsville
  - Princess Alexandra Hospital, Woolloongabba
- Austria (5):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Landesklinikum Krems, Krems
  - Kepler University Hospital, Linz
  - Wiener Gesundheitsverband Klinik Penzing, Vienna
  - Klinik Floridsdorf, Vienna
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Jessa Ziekenhuis Hospital, Hasselt
  - Centre Hospitalier Universitaire de Liege, Liège
  - AZ DELTA, Roeselare
  - Chu Ucl Namur, Yvoir
- Brazil (11):
  - Departmento de Pesquisa Clinica- Hospital de Amor de Barretos, Barretos
  - Cepon - Centro de Pesquisas Oncolăgicas de Santa Catarina, Florianópolis
  - Clínica de Neoplasias Litoral, Itajaí
  - Hospital São Lucas Da Pucrs, Porto Alegre
  - Cepho Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
  - ICESP Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
  - Hospital Sirio-Libanes, São Paulo
  - Hospital Beneficăncia Portuguesa de Săo Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - A. C. Camargo Cancer Center, São Paulo
- Canada (5):
  - William Osler Health System - Brampton Civic Hospital, Brampton
  - Cross Cancer Institute, Edmonton
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
  - Princess Margaret Cancer Center, Toronto
  - Cancercare Manitoba, Winnipeg
- China (26):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital,Capital Medical University, Beijing
  - Jilin Province Tumor Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Harbin Medical University Cancer Hospital, Haerbin
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliated Hospital of Nanchang University, Jiangxi
  - Shandong Cancer Hospital, Jinan
  - Linyi Cancer Hospital, Linyi
  - The Second Peoples Hospital of Neijiang, Neijiang
  - Yantai Yuhuangding Hospital, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Huazhong University of Science and Technology - Tongji Medical College - Tongji Hospital Tjh, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xiân Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Krajska Nemocnice Liberec A.S., Liberec
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni Thomayerova Nemocnice, Prague
- France (17):
  - Institut Sainte Catherine, Avignon
  - Chu Bordeaux, Bordeaux
  - Centre Hospitalier Intercommunal de Crăteil, Créteil
  - Institut Cœur Poumon CHU de Lille, Lille
  - Chu Limoges - Hopital Du Cluzeau, Limoges
  - Centre Léon Bérard, Lyon
  - Assistance Publique-Hăpitaux de Marseille, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Institut Régional Du Cancer de Montpellier, Montpellier
  - Ch de Mulhouse - Hăpital Emile Muller, Mulhouse
  - Institut Curie - Site de Paris, Paris
  - Hopital Tenon, Paris
  - Chu Rennes - Hopital Pontchaillou, Rennes
  - Chu Nantes - Hăpital Guillaume Et Renă Laănnec, Saint-Herblain
  - Institut de Cancerologie de La Loire, Saint-Priest-en-Jarez
  - Hăpital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (14):
  - Evangelische Lungenklinik Berlin, Berlin
  - Helios Klinikum Erfurt, Erfurt
  - Universtitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest Gmbh, Frankfurt
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting
  - Srh Wald-Klinikum Gera Gmbh, Gera
  - UNIVERSITATSKLINIKUM GIeBEN UND MARBURG GMBH, Giessen
  - Asklepios Klinik Harburg, Hamburg
  - Lki Lungenfachklinik Immenhausen, Immenhausen
  - Staedtisches Krankenhaus Kiel, Kiel
  - Johannes Wesling Klinikum Minden, Minden
  - Pius-Hospital Oldenburg, Oldenburg
  - Universitaetsklinikum Ulm, Ulm
- Greece (8):
  - 'Henry Dynant' Hospital Center, Athens
  - General Hospital of Athens of Chest Diseases 'Sotiria', Athens
  - General Hospital of Athens Alexandra, Athens
  - University General Hospital "Attikon", Chaïdári
  - University General Hospital of Larissa, Larissa
  - General Hospital of Patra Agios Andreas, Pátrai
  - Metropolitan Hospital, Piraeus
  - St Luke'S Hospital, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
- Italy (16):
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Humanitas Gavazzeni, Bergamo
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Universitaria Policlinico - Vittorio Emanuele (Presidio Gaspare Rodolico), Catania
  - Azienda Ospedaliero Universitaria Renato Dulbecco, Catanzaro
  - Istituto Nazionale Per La Ricerca Sul Cancro Di Genova, Genova
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Di Monza (Presidio San Gerardo), Monza
  - Azienda Ospedaliera Universitaria- Universită Degli Studi Della Campania Âluigi Vanvitelliâ, Napoli
  - Azienda Ospedaliero Universitaria Di Parma, Parma
  - Azienda Ospedaliera Di Perugia Ospedale S. Maria Della Misericordia, Perugia
  - Istituto Nazionale Tumori Regina Elena Irccs, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Centro Ricerche Cliniche Di Verona S.R.L., Verona
- Japan (13):
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Kansai Medical University Hospital, Hirakata-shi
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nakatogari
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osaka-Sakai
  - Kitasato University Hospital, Sagamihara
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Netherlands Cancer Institute, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Etz Elisabeth, Tilburg
- Poland (5):
  - Centrum Onkologii Im. Prof. F. Lukaszczyka W Bydgoszczy, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Szpital Specjalistyczny W Prabutach, Prabuty
  - Provita Prolife, Tomaszów Mazowiecki
- Portugal (5):
  - Centro Hospitalar E Universitărio de Coimbra E.P.E., Coimbra
  - Hospital Da Senhora Da Oliveira Guimarăes, Guimarães
  - Hospital Da Luz, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar Do Porto, E.P.E. - Hospital de Santo António, Porto
- Romania (4):
  - S.C Radiotherapy Center Cluj S.R.L, Bucharest
  - Institutul Oncologic 'Prof. Dr. Ion Chiricuta' Cluj Napoca, Cluj-Napoca
  - S.C Centrul de Oncologie Sfantul Nectarie Craiova, Craiova
  - S.C. Sigmedical Services Srl, Suceava
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent'S Hospital, Suwon
  - Ajou University Hospital, Suwon
- Spain (17):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Hospital de Especialidades de Jerez de La Frontera, Jerez de la Frontera
  - Ico L'Hospitalet - Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville
- Switzerland (3):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hfr Fribourg/Kantonsspital Fribourg, Villars-sur-Glâne
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospitalx, Tainan
  - National Taiwan University Cancer Centre, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- Turkey (Türkiye) (7):
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Dicle University, Medical Faculty, Diyarbakır
  - Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Izmir Medicalpark Hospital, Izmir
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - St James'S University Hospital, Leeds
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Owonikoko TK, Byers L, Cheng Y, Hayashi H, Paz-Ares L, Perol M, Hu H, Qian M, Garcia CR, Godard J, Tang M, Rudin CM. IDeate-Lung02: a Phase 3 study of second-line ifinatamab deruxtecan in patients with relapsed small cell lung cancer. Future Oncol. 2025 Oct;21(25):3275-3282. doi: 10.1080/14796694.2025.2565995. Epub 2025 Oct 7. PMID 41055143